CLINICAL TRIAL: NCT04007302
Title: Modification de l'activité du Cortex préfrontal Induite Par Distraction en réalité Virtuelle Chez le Sujet Lombalgique Chronique.
Brief Title: Modification of the Activity of the Prefrontal Cortex by Virtual Distraction in the Lumbago
Acronym: NGUYEN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: LOCAL 2017/DMNG-01; 2017-A02958-45 (Other: ANSM, France)
Record Dates: First submitted 2019-07-01; First posted 2019-07-05 (Actual); Last update posted 2019-07-08 (Actual); Status verified 2019-07

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — Spectroscopy, Near-Infrared

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- walking with distraction (Experimental): the patient walks in front of a screen with virtual reality simulation
  Interventions: Other: measurement of bilateral activity of the prefrontal cortex by a NIRS system (near infrared spectroscopy); Other: completion of questionnaires; Other: completion of questionnaires for pain
- Walking without distraction (Active Comparator): the patient walks on a treadmill without virtual reality simulation
  Interventions: Other: measurement of bilateral activity of the prefrontal cortex by a NIRS system (near infrared spectroscopy); Other: completion of questionnaires; Other: completion of questionnaires for pain

INTERVENTIONS:
Other: measurement of bilateral activity of the prefrontal cortex by a NIRS system (near infrared spectroscopy) — measurement of the cerebral oxygenation response by the use of the Near Infrared Spectroscopy (NIRS) method
Other: completion of questionnaires — igroup presence questionnaire (IPQ), Dallas Pain Questionnaire (DRAD), Fear-Avoidance Beliefs (FABQ) and Quebec Back Lumbago Scale
Other: completion of questionnaires for pain — analogical visual and numerical scale and Borg scale

SUMMARY:
The hypothesis of this work is that distraction is an effective way to modify the feeling and experience of chronic lumbar pain by modifying the functioning of the prefrontal cortex.

The main objective of this study is to show that during chronic low back pain generated during physical exercise, virtual reality distraction leads to the modification of the activity of the prefrontal cortex.

The secondary objectives are:

* Show a significant decrease in the average pain assessed with EVA during physical exercise with virtual reality distraction.
* Show an increase in the distance travelled with virtual reality distraction.
* Observe a decrease in perceived effort with virtual reality distraction.
* Quantify the adherence (presence) of subjects to the virtual environment

DETAILED DESCRIPTION:
A pre-test phase at D0 will be carried out with the objective of individually determining the exercise conditions (speed and slope) of walking that will generate lumbar pain. Patients who have not experienced lumbar pain during this phase will be excluded from the study. The patients included are then randomized according to the order of physical exercise situations.

For the tests, patients will be equipped with a miniaturized wireless (Octamon, Artinis) and multi-channel (8 optodes) NIRS device placed on the patient's frontal lobe according to EEG 10-20 positioning (fig. 2). They will then be placed on an inclined treadmill according to the angle that caused the pain during the pre-test.

During the test, subjects will walk to the voluntary stop and the different reasons for the stop (feeling of fatigue, pain, etc.) will be recorded by visual analogue scales and questionnaires. The duration of the exercise will be measured by a digital stopwatch connected to the treadmill. During physical exercise, the bilateral activity of the prefrontal cortex will be recorded continuously at a sampling frequency of 10 Hz.

For each test, subjects will be confronted with 2 situations, on D1 and D2. In a situation, walking will be done without distraction. In the other situation, the patient will be placed in front of a screen with virtual reality simulation while performing the walking exercise.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given free and informed consent and signed the consent
* The patient must be a member or beneficiary of a health insurance plan
* The patient is available for a 3-day follow-up
* The patient is between 18 and 75 years old
* Disabling lumbar pain beyond three months

Exclusion Criteria:

* Subject participates in another intervention study
* Subject is in an exclusion period determined by a previous study
* The subject is under the protection of justice, guardianship or curatorship
* Subject refuses to sign consent
* It is impossible to provide informed information about the subject
* The subject is unable to complete the study questionnaires
* The patient is pregnant, parturient, or breastfeeding
* The subject has a contraindication (or incompatible drug combination) for a treatment required for this study
* Recent involuntary weight loss
* Inflammatory schedule pain (predominantly nocturnal, requiring early morning rusting, improved by physical activity)
* Associated fever,
* Saddle anaesthesia
* Vesico-sphincterial disorders
* Typical root symptoms
* Systemic corticosteroid therapy
* History of cancer
* History of spinal trauma
* History of intravenous drug use
* Systemic corticosteroid therapy
* Surgical intervention of the spine or lower limbs
* Painful pathology of the lower limbs (coxarthrosis, gonarthrosis, vascular claudication or neurogenic when walking).

Exclusion criteria:

● Taking prescribed analgesic treatment after the inclusion procedure.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-09-09 (Actual); Primary Completion 2018-11-03 (Actual); Study Completion 2018-11-03 (Actual)

PRIMARY OUTCOMES:
measurement of prefrontal cortex activity | Day 1
  Brain oxygenation responses will be measured by the use of the Near Infrared Spectroscopy (NIRS) method (µmolar*cm)
measurement of prefrontal cortex activity | Day 2
  Brain oxygenation responses will be measured by the use of the Near Infrared Spectroscopy (NIRS) method (µmolar*cm)

SECONDARY OUTCOMES:
assessment of average pain | Inclusion
  analogical visual and numerical scale (0, no pain - 10 max pain)
assessment of average pain | Day 1
  analogical visual and numerical scale (0, no pain - 10 max pain)
assessment of average pain | Day 2
  analogical visual and numerical scale (0, no pain - 10 max pain)
measurement of the distance travelled | Inclusion
  meters
measurement of the distance travelled | Day 1
  meters
measurement of the distance travelleddistraction. | Day 2
  meters
Observe a decrease in perceived effort with virtual reality distraction. | Inclusion
  Borg's scale (0-10)
measurement of perceived effort | Day 1
  Borg's scale (0-10)
measurement of perceived effort | Day 2
  Borg's scale (0-10)
measurement of perceived effort | Day 1
  IPQ questionary (-3 ; +3)
Quantify patients' adherence (presence) to the virtual environment | Day 2
  IPQ questionary (-3 ; +3)

CONTACTS AND LOCATIONS:
Overall Officials: Anissa MEGZARI, Study Director — Centre Hospitalier Universitaire de Nīmes
Locations (1):
- CHU de Nîmes, Nîmes, France

IPD SHARING:
Plan to Share IPD: No